CLINICAL TRIAL: NCT01063114
Title: Proton Beam Radiotherapy for Medulloblastoma and Pineoblastoma: An Assessment of Acute Toxicity and Long Term Neurocognitive, Neuroendocrine and Ototoxicity Outcomes
Brief Title: Proton Beam Radiotherapy for Medulloblastoma and Pineoblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Torunn Yock, MD, Director, Pediatric Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-361; P01CA021239 (NIH)
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Brain Tumor; Medulloblastoma; Pineoblastoma
Keywords: proton beam radiation
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Pinealoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Beam Radiation (Experimental): Proton Beam Radiation
  Interventions: Radiation: proton beam radiation

INTERVENTIONS:
Radiation: proton beam radiation — Given once a day, 5 days a week (Monday-Friday)

SUMMARY:
There are two types of external radiation treatments (proton beam and photon beam). As part of the participant's treatment, they will receive radiation to the entire central nervous system (CNS); this is known as craniospinal irradiation (CSI). In the past, photon radiation therapy has been used for CSI. In this study we will be examining the effects of proton beam radiation therapy. Studies have suggested that this kind of radiation can cause less damage to normal tissue than photon radiation therapy. The physical characteristics of proton beam radiation let the doctor safely deliver the amount of radiation delivered to the tumor that is normally delivered through standard therapy but spare more normal tissue in the process.

DETAILED DESCRIPTION:
* Before beginning radiation therapy, participants will have scans done in order to prepare for the radiation treatment. Doctors will use information gathered from these scans to plan the best way to deliver radiation to the tumor.
* The following procedures will be performed either before or during the radiotherapy: Hearing exam; neurocognitive exam; blood tests and cerebral spinal fluid test.
* Not everyone who participates in this study will receive the same amount of proton radiation therapy. The length of time and amount of radiation received will depend upon the condition of the participant's disease. Radiation treatment will be given once a day, 5 days a week (Monday-Friday). The overall treatment course will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have undergone biopsy or attempted surgical resection and must have histologically confirmed medulloblastoma or pineoblastoma.
* Participants may have had a gross total resection, sub-total resection or biopsy only.
* For patients with no prior chemotherapy, treatment must start within 35 days of definitive surgery or as indicated if enrolled on therapeutic study
* Age range between 3 and 25 at the time of enrollment
* Life expectancy of greater than 3 months
* Blood laboratory values as outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Patients with more than one previous chemotherapy regimen
* Patients with recurrent or progressive disease after one or more regimens of pre-radiation chemotherapy
* Patients with prior radiation therapy
* Any major uncontrolled or poorly controlled intercurrent illness that would limit compliance with study requirements
* Pregnant women

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04-08 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torunn I Yock, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Vatner RE, Niemierko A, Misra M, Weyman EA, Goebel CP, Ebb DH, Jones RM, Huang MS, Mahajan A, Grosshans DR, Paulino AC, Stanley T, MacDonald SM, Tarbell NJ, Yock TI. Endocrine Deficiency As a Function of Radiation Dose to the Hypothalamus and Pituitary in Pediatric and Young Adult Patients With Brain Tumors. J Clin Oncol. 2018 Oct 1;36(28):2854-2862. doi: 10.1200/JCO.2018.78.1492. Epub 2018 Aug 17. PMID 30118397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Beam Radiation
Started | 90
Completed | 89
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.3 [6.4 to 12.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 79
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Ototoxicity
Description: Cumulative incidence (estimated percentage participants) who experienced ototoxicity defined as either grade 3 or 4 hearing loss in either ear after the completion of radiation therapy in the overall participant population. Cumulative incidence and 95% confidence intervals are shown at 3- and 5-years post RT (radiation treatment)
Time Frame: 3- and 5- years post radiation treatment
Population: Subset of study population that were at risk of developing a grade 3 or 4 hearing loss in either ear in follow-up after the completion of radiation therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 77
percentage of participants
  3-Years post RT (radiation treatment) | 26 [16 to 37]
  5-Years post RT | 27 [17 to 38]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; 3-Year Cumulative incidence = 26, 95% CI 2-sided [16 to 37]
Statistical Analysis 2: Comparison: Proton Beam Radiation; Test type: Other; 5-Year Cumulative incidence = 27, 95% CI 2-sided [17 to 38]

2. Primary Outcome: Endocrine Dysfunction
Description: Cumulative incidence (estimated percentage participants) that developed endocrine dysfunction at 3- and 5-years following completion of proton radiation therapy.
Time Frame: 3- and 5- years post radiation treatment
Population: Patient population at risk of developing an endocrine dysfunction during follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 90
percentage of participants
  3-Years post RT | 46 [34 to 57]
  5-Years post RT | 67 [54 to 77]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; 3-Year Cumulative incidence = 46, 95% CI 2-sided [34 to 57]
Statistical Analysis 2: Comparison: Proton Beam Radiation; Test type: Other; 5-Year Cumulative incidence = 67, 95% CI 2-sided [54 to 77]

3. Primary Outcome: Neurocognitive Effects
Description: Difference in Full-Scale Intelligence Quotient (FSIQ) between baseline and latest follow-up neurocognitive test. Tests used include WISC (Wechsler Intelligence Scale for Children) IV, WISC V, WAIS (Wechsler Adult Intelligence Scale) III, WAIS IV. The test measures the FSIQ of children through four indices; the Verbal Comprehension Index (VCI), Perceptual Reasoning Index (PRI), working memory test, and a processing speed test. FSIQ and the four indices are all assessed on a bell curve scale with an average score of 100 and standard deviation of 15. Higher scores represent higher intelligence and lower scores represent reduced intelligence.
Time Frame: Baseline and Follow-up (median of 6 years)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 26
score on a scale
  Baseline FSIQ | 102.7 (12.5)
  Follow-up FSIQ | 91.7 (20.5)
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; p = 0.01024, t-test, 2 sided; Paired t test; Mean Difference (Net) = -11.0, 95% CI 2-sided [-19.2 to -2.9]

4. Secondary Outcome: Progression Free Survival
Description: 3- and 5-year progression free survival rate of pediatric medulloblastoma and pineoblastoma patients treated with proton CSI treatment.
Time Frame: 3- and 5-years post radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 90
percentage of participants
  3-Year post RT | 83.2 [75.8 to 91.3]
  5-Year post RT | 79.6 [71.7 to 88.5]
Statistical Analysis 1: Comparison: Proton Beam Radiation; Test type: Other; 3-Year Survival Probability = 83.2, 95% CI 2-sided [75.8 to 91.3]
Statistical Analysis 2: Comparison: Proton Beam Radiation; Test type: Other; 5-Year Survival Probability = 79.6, 95% CI 2-sided [71.7 to 88.5]

5. Secondary Outcome: Treatment Efficiency
Description: To modify the speed of treating patients requiring cranial spinal irradiation (CSI) and improve the safety of treating patients under anesthesia
Time Frame: 2 years
Population: It was not possible to change/alter any portion of the treatment process for those requiring CSI and therefore no patient had altered treatment times. Specifically, we were unable to speed the delivery of the radiation and make treatment scheduling slots shorter than they already were. With no changes in treatment speed across patients, potential outcomes in terms of safety and treatment efficiency could not be compared by treatment speed. This data will not be collected in the future.
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Who Experienced an Acute Toxicity by Grade
Description: All patients shall be assessed for acute toxicity on a weekly basis during craniospinal irradiation (CSI). Percentage of participants who experienced an acute toxicity by grade. Acute toxicities are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Toxicities are graded on a scale of 1 to 5. A higher grade indicates a worse outcome with 1 being mild, 4 being life-threatening, and 5 being death.
Time Frame: 3 months after radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Beam Radiation
Number analyzed (Participants) | 90
Participants
  Grade 1 | 90
  Grade 2 | 84
  Grade 3 | 36
  Grade 4 | 12
  Grade 5 | 0

ADVERSE EVENTS:
Time Frame: Through start of radiotherapy treatment to study end (up to 5 years post radiation treatment)
Description: All adverse events experienced by participants will be collected from the time of the first dose of study treatment, through the study and until the final study visit. All patients were assessed for acute toxicity on a weekly basis during CSI. Grading of acute toxicity was done per the CTEP (Cancer Therapy Evaluation Program) Active Version of CTCAE (Common Terminology Criteria for Adverse Events).
Arm/Group | Proton Beam Radiation
All-Cause Mortality (participants affected / at risk) | 19/90
Serious Adverse Events (participants affected / at risk) | 9/90
Other Adverse Events (participants affected / at risk) | 89/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=90)
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anemia (Blood and lymphatic system disorders) | 3
Middle ear inflammation (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Eye infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
Neutrophil count decreased (Investigations) | 4
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proton Beam Radiation (N=90)
Abdominal pain (Gastrointestinal disorders) | 4
Agitation (Psychiatric disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 81
Anemia (Blood and lymphatic system disorders) | 24
Anorexia (Metabolism and nutrition disorders) | 56
Anxiety (Psychiatric disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
CD4 lymphocytes decreased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 79
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 7
Dry eye (Eye disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 10
Dysesthesia (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 4
Ear pain (Ear and labyrinth disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 7
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 6
External ear inflammation (Ear and labyrinth disorders) | 2
Fatigue (General disorders) | 72
Gait disturbance (General disorders) | 3
Growth suppression (Musculoskeletal and connective tissue disorders) | 29
Headache (Nervous system disorders) | 40
Hearing impaired (Ear and labyrinth disorders) | 48
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 4
Lymphocyte count decreased (Investigations) | 27
Mucosal infection (Infections and infestations) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 60
Neutrophil count decreased (Investigations) | 25
Pain (General disorders) | 5
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Photophobia (Eye disorders) | 1
Platelet count decreased (Investigations) | 19
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 22
Sore throat (Respiratory, thoracic and mediastinal disorders) | 27
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 51
Weight loss (Investigations) | 32
White blood cell decreased (Investigations) | 32
Tinnitus (Ear and labyrinth disorders) | 3
Precocious puberty (Endocrine disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 10
Delayed puberty (Endocrine disorders) | 3
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 16
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 7
Fever (General disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Blood gonadotrophin abnormal (Investigations) | 4
Blood prolactin abnormal (Investigations) | 2
Growth hormone abnormal (Investigations) | 25
Weight gain (Investigations) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 7
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acoustic nerve disorder NOS (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 7
Central nervous system necrosis (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 34
Concentration impairment (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
IVth nerve disorder (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 4
Nystagmus (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 6
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT01063114/Prot_SAP_000.pdf